CLINICAL TRIAL: NCT07003529
Title: Rôle Des Colliculi inférieurs Dans Les Hallucinations Auditives : étude Pilote Par Neuroimagerie
Brief Title: Role of Inferior Colliculi in Auditory Hallucinations
Acronym: SchizoHIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NIMAO2024-2/MP-01
Record Dates: First submitted 2025-05-20; First posted 2025-06-04 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia; Hallucinations, Auditory
MeSH Terms: conditions — Schizophrenia; Hallucinations

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Group (SCZ+/AH+) (Experimental): schizophrenic patients experiencing auditory hallucinations
  Interventions: Other: Unenhanced brain MRI
- Control Group (SCZ+/AH-) (Experimental): schizophrenic patients without hallucinations
  Interventions: Other: Unenhanced brain MRI

INTERVENTIONS:
Other: Unenhanced brain MRI — Unenhanced brain MRI in five sequences: 1) T1-weighted anatomical sequences 2) Resting-state functional sequences 3) Task-based functional sequence 4) Structural sequence using Diffusion Tensor Imaging (DTI) 5) Routine magnetic resonance spectroscopy sequence

SUMMARY:
The neural basis of auditory hallucinations (AH) in patients with schizophrenia is poorly characterized. Functional imaging studies investigate either the "state" dimension (i.e., the measurement of changes in brain area activation at the precise moment of AH onset) or the "trait" dimension (i.e., the neural correlates of the propensity to hallucinate). A corollary of AH (particularly acoustic-verbal) is the activation of brain regions involved in the auditory perception of speech (auditory cortex). One theory is that patients with schizophrenia with AH may have a deficit in processing their internal speech (i.e., external attribution to internal verbal content). However, there is little clinical data on the specific role of the mesencephalic region of the inferior colliculi (IC) in the formation of these symptoms. Preliminary research has shown intense expression of dopamine D2 receptors, particularly on glutamatergic neurons in mouse ICs. Thus, ICs receive numerous inhibitory dopaminergic inputs, likely involved in signal optimization and modulation. The study authors hypothesize that AHs are the result of a defect in signal inhibition by the IC, which lose their function as perceptual filters.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* DSM-5 diagnosis of schizophrenic disorder (based on clinical assessment and confirmed by the MINI 7.0 interview)
* Patient with a schizophrenic disorder lasting ≤ 20 years
* Patient treated in a psychiatric unit as an inpatient (in non-specialized care) or outpatient or under a mandatory ambulatory psychiatric care programme
* Clinical condition compatible with imaging based on clinical judgment
* Ability to understand, write, and read French

Specific inclusion criteria for the group (SCZ+/HA+) • Patient with a PANSS score (question P3 regarding hallucinations) ≥ 4 (corresponds to PANSS (P3) 4, 5, 6, and 7 patients) AND having experienced hallucinations in the past 15 days.

Specific inclusion criteria for the control group

• Patient with a PANSS score (question P3 regarding hallucinations) = 1) AND having not experienced any hallucinations in the past 15 days.

Exclusion Criteria:

* The patient is under safeguard of justice or state guardianship
* Contraindications to magnetic resonance imaging, including severe claustrophobia, based on clinical judgment.
* Congenital or acquired deafness
* Suicide risk, based on clinical judgment
* Patient with moderate to severe intellectual disability, based on medical records
* Patient with moderate to severe neurocognitive disorders, based on medical records
* Patient receiving anticholinergic therapy (biperiden-Akineton, trihexyphenidyl-Artane, tropatepine-Lepticur)
* Patient participating in an interventional study involving a drug or medical device, or a Category 1 RIPH within 3 months prior to inclusion
* Person under judicial protection
* Pregnant, parturient, or breastfeeding woman
* Person unable to express consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Resting state of functional connectivity of the inferior colliculi region with other regions of the auditory network between groups | Day 0
  Measured by MRI
Default mode network patterns between groups | Day 0
  Measured by MRI

SECONDARY OUTCOMES:
Neuronal activation in the ICs during exposure to auditory stimuli between groups | Day 0
  Difference in the blood-oxygen level dependent (BOLD) signal measured by functional MRI during an auditory stimulus exposure paradigm in the IC region
Per-auditory activation in other brain areas between groups | Day 0
  Difference in the BOLD signal measured by functional MRI in other brain areas
IC metabolite composition between the groups | Day 0
  Difference in the peak magnetic resonance spectrometry (sMRI) signal
Structural connectivity via white matter between ICs and other auditory network structures between groups | Day 0
  Difference in structural connectivity using DTI (diffusion tensor imaging, anisotropy fraction calculation, mean diffusivity, and tractography) from the ICs
Correlation between BOLD signal and psychopathological symptoms | Day 0
  Measured by Positive and Negative Syndrome Scale (PANSS), providing a negative symptomatology score ranging from 7 to 49, and a general psychopathology score ranging from 16 to 112, with a total score ranging from 30 to 210.
Correlation between BOLD signal and severity of delusions and hallucinations | Day 0
  Measured by Psychotic Symptom Rating Scale (PSYRATS), an 11-item scale where each symptom is rated from 0 to 4 depending on the intensity
Correlation between BOLD signal and doses of antipsychotic treatment | Day 0
  Antipsychotic doses calculated by olanzapine equivalent method
Difference in perauditory activation and functional connectivity (resting-state) in SCZ+ HA+ patients who hallucinated during the procedure and those who did not | Day 0
  Measured via post-hoc task-based, BOLD signal state hallucination analysis
Correlation between BOLD signal and dissociation symptoms | Day 0
  Measured by Dissociative Experience Scale (DES)
Correlation between BOLD signal and severity of somatoform manifestations of dissociation | Day 0
  Measured by Somatoform Dissociation Questionnaire (SDQ)
Correlation between BOLD signal and clinically assessed states of dissociation | Day 0
  Measured by Clinician Administered Dissociative States Scale (CADSS), a 5-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Martin Pastre, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nîmes, Hôpital Universitaire Carémeau, Nîmes, France